CLINICAL TRIAL: NCT07342036
Title: Prospective Study of Lead-associated Tricuspid Regurgitation in Patients Undergoing New Transvalvular Lead Insertion
Acronym: LITR
Status: Recruiting | Type: Observational
Sponsor: Hazem Omran (Other)
Responsible Party: Sponsor-Investigator, Hazem Omran, Attending Physician, Clinic for General and Interventional Cardiology/Angiology, Herz- und Diabeteszentrum NRW
Organization: Clinic for General and Interventional Cardiology/Angiology, Herz- und Diabeteszentrum NRW (Other)
Other Study IDs: HDZ-KA_024_HO
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Tricuspid Valve Regurgitation; Pacemaker; ICD; Left Bundle Branch Area Pacing
Keywords: tricuspid regurgitation; lead-related TR; lead-associated TR
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pacemaker-standard: Only pacemaker with standard positioning (no ICD leads, no LBBaP)
- ICD: any ICD leads through tricuspid valve
- LBBaP: Left bundle branch area pacing leads

SUMMARY:
The goal of this clinical trial is to record the incidence of newly developed or worsening tricuspid valve regurgitation (TR) following the implantation of a pacemaker or defibrillator with a transvenous lead. To collect this data, a transthoracic echocardiogram (TTE) with 3D imaging of the tricuspid valve (TV) will be performed before and after pacemaker implantation, with particular emphasis on assessing the tricuspid valve. Additionally, routine follow-up visits will be conducted at 6 and 12 months post-intervention, during which a TTE, ECG, NT-proBNP measurement, and pacemaker check will be performed.

DETAILED DESCRIPTION:
The prevalence of tricuspid regurgitation (TR) in patients with a pacemaker or ICD/CRT device varies widely, ranging from 5% to 45% across different study protocols. To date, only retrospective analyses have shown that implantation of a device with a transvalvular lead can cause or worsen TR, highlighting the importance of early diagnosis. The aim of this study is to prospectively evaluate patients indicated for cardiac electronic device implantation to document the incidence of newly developed regurgitation (greater than trace) or worsening of existing regurgitation (by at least one grade). Additionally, the study will investigate predictive factors for the development or progression of TR.

ELIGIBILITY:
Inclusion Criteria:

* medically indicated for pacemaker, ICD- or CRT implantation
* No previous diagnosis of severe tricuspid regurgitation on enrollment
* No existing transvalvular device (must be first implantation)
* No other diagnosed severe valvular heart disease
* Not previous diagnosis with pre-capillary pulmonary hypertension
* No previous diagnosis of structural disease of the right ventricle (i.e. ACM, cardiac sarcoidosis, carcinoid...)

Exclusion Criteria:

* Patients unable to give consent
* Under the age of 18 years
* Relevant pre-capillary pulmonary hypertension according to decision of the heart-team (sPAP echo >70 mmHg)
* Severe tricuspid valve regurgitation (Grade 3 or worse) on enrollment
* Patients who have undergone Lead-explantation
* Exisiting valvular heart disease requiring treatment according to the decision of the heart-team. These patients may be enrolled in the study following treatment.
* Previous tricuspid valve surgery
* Patients with congenital heart disease (i.e. tetralogy of fallot, Ebstein's anomaly,...)
* Pregnant or breastfeeding women
* Life expectancy < 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have been indicated to have a new cardiac device with a transvalvular probe implanted for any given indication
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Worsening of TR of at least 1 grade | over the sutdy period up to 1 year after lead insertion
  Worsening of tricuspid regurgitation of at least one grade from baseline before lead insertion through tricuspid valve

SECONDARY OUTCOMES:
TR > mild at follow-up | during study time frame up to 1 year after Pacemaker/ICD implantation
  The percentage of patients with at least moderate TR or worse
NTproBNP change from baseline | at 6 and at 12 months after Pacemaker/ICD implantation
  Change in NTproBNP levels from baseline to 6 and 12 Months
Hospitalization for heart failure (HFH) | up to 12 months after Pacemaker/ICD implantation
  Any uplanned hopsitalization with requirement of iv diuretics therapy after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Hazem Omran, MD, Principal Investigator — Herz- und Diabeteszentrum NRW
Locations (1):
- Herz- und Diabeteszentrum NRW, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No